CLINICAL TRIAL: NCT04379063
Title: COVID-19 Pandemic Short Interval National Survey Gauging Psychological Distress Among Physicians (COPING Survey): A Longitudinal Survey
Brief Title: COVID-19 Pandemic Short Interval National Survey Gauging Psychological Distress
Acronym: COPING
Status: Completed | Type: Observational
Sponsor: Jon Bailey (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Jon Bailey, Anesthesiolgist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Other Study IDs: NSHA REB#1025690
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Burnout, Professional; Psychological Distress
Keywords: COVID-19; Coronavirus; Pandemic; Outbreak
MeSH Terms: conditions — Burnout, Professional; COVID-19; Coronavirus Infections | interventions — Pandemic Preparedness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Canadian physicians during COVID-19 pandemic: Any physician who is practicing in Canada during the COVID-19 pandemic, whether they hold a full, provisional, or post-graduate in-training license.
  Interventions: Other: COVID-19 pandemic

INTERVENTIONS:
Other: COVID-19 pandemic — Currently practicing during the COVID-19 pandemic

SUMMARY:
The Coronavirus Disease (COVID-19) pandemic is unprecedented in its scale of infection and the response required to decrease the mortality rates. Disturbingly, the European and United States experience demonstrates that health care systems in industrialized countries are at risk of becoming overwhelmed. Physicians are already at risk of burnout under normal working conditions, and in particular, when responding to crisis situations. During the 2003 severe acute respiratory syndrome (SARS) outbreak, healthcare workers experienced high rates of psychological distress that lasted years. However, there may be protective factors that may decrease the rate or severity of psychological distress and burnout. This study seeks to investigate the rates of physician burnout assessed at multiple time points during the COVID-19 pandemic. Further, this study seeks to determine the factors that may increase or decrease burnout and psychological distress in such a setting.

This study will be a national longitudinal survey of physicians in Canada. It will include all physicians that currently hold a license to practice in Canada (whether in training or a full license). Consenting participants will complete an initial survey gathering information about their type of practice, health conditions, preparations the COVID-19 pandemic, burnout, and psychological distress. Every month, participants will be asked to complete a follow-up survey, describing their stressors, coping strategies, burnout, and psychological distress.

The investigators will analyze and report the initial results to help provincial and national organizations support our physicians and mitigate burnout during this pandemic. The results of the follow up surveys will be analyzed and reported following the pandemic. These findings will help keep our physician workforce healthy under normal working conditions and during future crises.

DETAILED DESCRIPTION:
Background It has become ubiquitous to describe the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pandemic and the global measures to decrease mortality rates of Coronavirus Disease (COVID-19) as 'unprecedented'. The Public Health Agency of Canada (PHAC) models released on April 8th predict that even with strict epidemiologic controls 934,000-1,879,000 people will be infected in Canada and 11,000- 22,000 will die. Disturbingly, the European and United States experience demonstrates that health care systems in industrialized countries are at risk of becoming overwhelmed. It has long been recognized that physicians are at risk for burnout, which can negatively affect their ability to care for patients, their colleagues and themselves. Infectious disease pandemics present many of the same challenges for physicians as natural disasters and mass casualty events, with the addition of a prolonged time frame, potential need for isolation away from family, and concern of becoming infected or infecting loved ones. During the 2003 severe acute respiratory syndrome (SARS) outbreak, 18-57% of health care workers (HCWs) experienced measurable psychological distress. Even 1-2 years following the SARS pandemic HCWs in Ontario experienced high levels of burnout (19-30%), psychological distress (30-45%), and PTSD symptoms (8-13%). Despite the overall high rates, there are several mitigating factors that may decrease the rate or severity of psychological distress and burnout.

Given that these studies generally measure burnout and psychological distress at one or two cross-sectional time points, it is difficult to tell how burnout develops over time. Additionally, the bulk of the studies assessed HCWs following natural disasters, which tend to present as a single time point with one large wave of patients. The current crisis is distinct in its sustained level of demand on HCWs with potential for multiple waves of patients or a sustained high number of patients outstripping the health care system resources for months at a time. This study seeks to investigate the rates of burnout assessed at multiple time points during the COVID-19 pandemic. Further, this study seeks to determine the relationship between patient numbers, mitigating factors, and exacerbating factors and the rates of burnout at various time points.

Objectives

1. What are the rates of psychological distress and burnout among physicians and residents throughout the COVID-19 pandemic?
2. What baseline factors are associated with reductions and increases in psychological distress and burnout over time (trajectories)?

Methods This study will be a national longitudinal survey of physicians in Canada. The sampling frame will be all physicians currently practicing in Canada, whether they hold a full, provisional, or post-graduate in-training license. The survey will be distributed by: 1. Advertisements on Twitter, 2. Provincial physician associations, and 3. National specialty groups for higher risk specialties (anesthesia, critical care, emergency medicine). Recipients will be directed to the survey site hosted by Redcap. Cross-sectional results of the initial survey to give immediate feedback to provincial and national organizations about the threat of physician burnout and psychological distress. Longitudinal results will analyze how burnout and distress change over time and will analyze the relationship to mitigating and exacerbating factors.

Consenting participants will complete an initial survey gathering demographic information (age, gender, trainee, years in practice, specialty, chronic health conditions, practice type (academic, community, rural), preparatory information (prior to first COVID-19 suspected case: COVID-19 pathways/procedures, simulation, designated areas, scheduling changes), and baseline measures (Maslach Burnout Inventory - General Survey (MBI-GS) short form, Pandemic Experience & Perceptions Scale (PEPS), Hospital Anxiety and Depression Scale (HADS), stressors, resources, coping strategies). Participants will then receive follow up questionnaires every month until there is a sustained period of no new cases in their province (1 month without a new case) up to a maximum of one-year involvement. These follow up questionnaires will measure burnout (MBI-GS), psychological distress (HADS), pandemic specific stressors (PEPS), workplace stressors, and resources/coping strategies. A final follow-up survey will be sought one year after the end of the short- interval surveys to assess the long-term effects of responding to the COVID pandemic.

Statistical Analysis Objective 1. Variables will be described using mean and standard deviation when normally distributed or median and interquartile range when skewed as measured by the Shapiro-Wilk test.

Objective 2. The cross-sectional results of the initial survey will be analyzed using linear regression to quantify the strength of relationship between factors and burnout. In the longitudinal analysis, trajectory analysis using latent growth mixed modelling (LGMM) will be used to identify trajectories of burnout and psychological distress amongst physicians over time. LGMM is ideally suited to longitudinal data as it is robust to the effects of missing data. Furthermore, LGMM may prove very useful in an unprecedented situation such as this in which there is scant data on which to base hypotheses as LGMM allows trajectories to be identified more empirically based on the data rather than through a priori conceptual models.

Anticipated Outcomes The investigators will discover whether the characteristics of burnout during this pandemic are comparable to the current body of knowledge about physician burnout at baseline or during more limited periods of crisis. This will inform whether current interventions for physician burnout are appropriate during widespread pandemic events, both as physicians continue to deal with COVID-19 and in the future. Improved understanding of stressors and protective factors will be essential not only for planning therapeutic studies at an individual level but will also allow institutions to mobilize high yield supports for physicians at risk.

ELIGIBILITY:
Inclusion Criteria:

* Any physician who is currently practicing in Canada, whether they hold a full, provisional, or post-graduate in-training license.

Exclusion Criteria:

* Non-physician healthcare providers, medical students, physicians without an active license to practice will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The membership of Canadian Medical Association (CMA) was 71,655 as of June 10, 2019. This includes medical students and retired physicians. The total number of residents (8,681) and practicing physicians (44,557) is 53,238 who could meet inclusion criteria. Response rates by medical trainees to web-based surveys without incentives are approximately 60%, based on previous survey studies. However, given the current situation and the potential for overwhelmed healthcare systems and personnel, we expect a much lower response rate of 20-30%.
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Burnout | Start of survey until there is a sustained period of no new cases in their province (1 month without a new case)
  Measured by the Maslach Burnout Inventory - General Survey (MBI-GS) short form. The MBI-SF has three subscales (exhaustion, cynicism, efficacy). Each subscale is scored from 0-6 indicating the frequency of work-related feelings. A higher score in both exhaustion and cynicism indicate burnout is more likely; whereas, higher scores in efficacy indicate burnout is less likely.
Psychological Distress | Start of survey until there is a sustained period of no new cases in their province (1 month without a new case)
  Measured by the Hospital Anxiety and Depression Scale (HADS). The HADS scores both symptoms of depression and anxiety using 14-item measure (7 item with possible scores 0-21 each). Higher scores suggest that depression and/or anxiety are more likely.

SECONDARY OUTCOMES:
Post-traumatic stress symptoms | One year following the end of the survey (no new cases in their province, 1 month without a new case)
  Measured by the Post-Traumatic Stress Disorder (PTSD) Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (PCL-5). Symptoms suggestive of PTSD are scored using a 20-item measure with possible scores ranging from 0-80. Higher scores are more suggestive of PTSD.
Post-traumatic growth | One year following the end of the survey (no new cases in their province, 1 month without a new case)
  Measured by the Post-traumatic Growth Inventory (PTGI-SF). The PTGI-SF is a 10-item measure with possible scores ranging from 0-50. Higher scores suggest that post-traumatic growth is more likely.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bailey JG, Wong M, Bailey K, Banfield JC, Barry G, Munro A, Kirkland S, Leiter M. Pandemic-related factors predicting physician burnout beyond established organizational factors: cross-sectional results from the COPING survey. Psychol Health Med. 2023 Jul-Dec;28(8):2353-2367. doi: 10.1080/13548506.2021.1990366. Epub 2021 Oct 14. PMID 34649468